CLINICAL TRIAL: NCT03915457
Title: Effects of Thigh Cuffs to Prevent the Deconditioning Induced by 5 Days of Dry Immersion Used as a Ground-based Model to Study the Effects of Weightlessness
Brief Title: Thigh Cuffs to Prevent the Deconditioning Induced by 5 Days of Dry Immersion
Acronym: DI-Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-179
Record Dates: First submitted 2019-03-05; First posted 2019-04-16 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-04

CONDITIONS: Weightlessness; Weightlessness; Adverse Effect
Keywords: Simulated Microgravity; Weightlessness; Countermeasure; Dry immersion; Supportlessness

STUDY DESIGN:
Intervention Model Description: A monocentric open parallel randomized and controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry immersion Control Group (Experimental): 5 days of dry-immersion
  Interventions: Other: Dry immersion Control Group
- Thigh Cuffs intervention (Experimental): 5 days of dry-immersion with thigh cuffs
  Interventions: Other: Thigh cuffs intervention

INTERVENTIONS:
Other: Dry immersion Control Group — Subjects are immersed up to the neck for 5 days in a specially designed bath filled with tap water.
  Arms: Dry immersion Control Group
Other: Thigh cuffs intervention — Subjects are immersed up to the neck for 5 days in a specially designed bath filled with tap water. During the 5 days of dry immersion, the subjects will wear the thigh cuffs daily for 10 hours during the day (8 am to 6 pm). Thigh cuffs are strips of fabric with inserts of elastic fabric. Different sizes exist to adapt to different thighs. Each cuff has five tightening positions (from 1 to 5) and they will be tightened at the upper third of the thighs to create an occlusion pressure of about 30 mmHg.
  Arms: Thigh Cuffs intervention

SUMMARY:
The objective of the study is to investigate whether thigh cuffs help to prevent and/or reduce the deconditioning induced by 5 days of dry immersion and in particular the fluid shift and its related ophthalmological disorders. During a randomized 5 day dry-immersion study in 20 healthy male adults the two following aims will be undertaken:

* Ten scientific protocols will assess the changes in the cerebral, ocular, cardiovascular, metabolism, cognitive, muscle and bone systems.
* In the above mentioned systems, the potential beneficial effects of the countermeasure protocol will also be investigated.

DETAILED DESCRIPTION:
Space flights have shown the possibilities and limitations of human adaptation to space. For the last 50 years, results showed that the space environment and microgravity in particular, cause changes that may affect the performance of astronauts. These physiological changes are now better known: prolonged exposure to a weightlessness environment can lead to significant loss of bone, muscle mass, strength, cardiovascular and sensory-motor deconditioning, immune, hormonal and metabolism changes. Nevertheless, more recent missions have revealed a new suite of physiological adaptations and consequences of space flight. Indeed, astronauts exposed to prolonged weightlessness experience hyperopic shifts and structural alteration in the eye (e.g., choroidal folds and optic disc edema). This condition was defined by NASA as Spaceflight-Associated Neuro-ocular Syndrome (SANS). Some of these vision changes remain unresolved for years after flight. This phenomenon has most likely existed since the beginning of human space flight, but is just recently being recognized as a major consequence of adaptation to microgravity. Changes in vision and eye structure are thought to be the result of prolonged exposure to space flight-induced headward fluid shifts and elevated intracranial pressure. Loss of the hydrostatic pressure gradient during spaceflight leads to this redistribution of body fluids toward the head. To prepare for future manned missions beyond the low Earth Orbit, the mechanisms underlying SANS syndrome have to be investigated and countermeasures designed to reverse or prevent SANS are required. Venoconstrictive thigh cuffs (VTCs) represent one possible countermeasure to mitigate a headward fluid shift. The Russian Space Agency uses VTCs (bracelets) to sequester fluid in the lower limbs and mitigate the subjective sensation of head congestion during space-flight. Moreover, experiments on 6-month Mir missions demonstrated that bracelets reduced jugular vein cross-sectional area in cosmonauts by 12% to 20%. However, it is unknown how VTCs (including bracelets) affect ocular physiologic features. The space agencies are actively engaged in studying the initiation and progression of SANS syndrome through studies on the International Space Station and on the ground. Indeed, considering the limited number of flight opportunities, the difficulties related to the performance of in-flight experiments (operational constraints for astronauts, limited capabilities of in-flight biomedical devices), ground-based experiments simulating the effects of weightlessness are used to better understand the mechanisms of physiological adaptation, design and validate the countermeasures. Different methods are used to simulate microgravity on Earth. However, two separate approaches, -6° head-down bed rest (HDBR) and dry immersion (DI) have provided possibilities for long-term exposures with findings closest to those seen with a weightless state. They produce changes in body composition (including body fluid redistribution), cardiovascular and skeletal muscle characteristics that resemble the effects of microgravity. The common physiological denominator is the combination of a cephalad shift of body fluids and reduced physical activity. Unlike bed rest, dry immersion provides a unique opportunity to study the physiological effects of the lack of a supporting structure for the body. Dry immersion means immersing into the thermoneutral water covered with special elastic free floating waterproof fabric. The subject, surrounded by film and "free suspended" in the water mass, remains dry. During horizontal immersion, pressure forces are distributed nearly equally around the entire surface of the body (only the head and neck are not entirely supported by water). The absence of mechanical support of specific zones during immersion creates a state akin to weightlessness that is called "supportlessness". Physiological changes under DI develop more rapidly and are more profound than under HDBR. This advanced ground-based model is extremely suited to test countermeasures for microgravity-induced deconditioning and physical inactivity-related pathologies.

The present study is organized in this context by the French space agency (CNES) to assess on twenty healthy male volunteers the effects of thigh cuffs to prevent the deconditioning induced by 5 days of dry immersion and in particular the fluid shift and its related ophthalmological disorders. Using an integrated approach, the CNES has selected ten scientific protocols to assess the changes in the different physiological fields and the potential beneficial effects of the countermeasure to prevent and/or reduce these changes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer (see below the description of medical tests and laboratory analysis performed at the selection visit),
* Age 20 to 45,
* No overweight nor excessive thinness with BMI (weight Kg/ height m2) between 20 and 26,
* Height between 158 and 185 cm,
* No personal nor family past record of chronic or acute disease or psychological disturbances which could affect the physiological data and/or create a risk for the subject during the experiment,
* Fitness level assessment:

  * if age < 35 years: 35 ml/min/kg < VO2max < 60ml/min/kg
  * if age > 35 years: 30 ml/min/kg < VO2max < 60ml/min/kg
* Walking between 7000 - 8000 steps/day,
* Active and free from any orthopedic (in particular no vertebral fracture, scoliosis or herniated disc) musculoskeletal and cardiovascular disorders,
* Non smokers,
* No alcohol, no drug dependence and no medical treatment,
* No antibiotic treatment in the 2 previous months before the beginning of the study,
* Covered by a Social Security system,
* Have signed the information consent,
* Free of any engagement during the study.

Exclusion Criteria:

* - Past record of orthostatic intolerance,
* Cardiac rhythm disorders,
* Chronic back pains,
* Vertebral fracture, scoliosis or herniated disc,
* Glaucoma,
* HTA,
* History of migraines,
* History of hiatus hernia or gastro-esophageal reflux,
* History of thyroid dysfunction, renal stones, diabetes,
* History of head trauma,
* Past records of thrombophlebitis, family history of thrombosis or positive response in thrombosis screening procedure (anti thrombin III, S-protein, C-protein, factor V Leiden mutation and the mutation 20210 of the prothrombin gene),
* Individuals exhibiting mutations involved in hereditary hemochromatosis (HAMP, HFE, HFE2, SCL40A1 and TRF2),
* Abnormal result for lower limbs echo-doppler,
* History or active claustrophobia,
* History of genetic muscle and bone diseases of any kind,
* Bone mineral density: T-score ≤ -1.5 on the hip,
* Osteosynthesis material, presence of metallic implants or any other contra-indication for MRI,
* Poor tolerance to blood sampling,
* Having given blood (more than 8ml/kg) in a period of 8 weeks or less before the start of the experiment,
* Antibiotic treatment in the 2 previous months before the beginning of the study,
* Vegetarian or vegan,
* History of food allergy,
* Positive reaction to any of the following tests: HVA IgM (hepatitis A), HBs antigen (hepatitis B), anti-HVC antibodies (hepatitis C), anti-HIV1+2 antibodies,
* Subject already participating or in the exclusion period of a clinical research,
* Refusal to give permission to contact his general practitioner,
* Incarcerated persons,
* Subject who, in the judgment of the investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject who has received more than 4500 Euros within 12 months for being a research subject.
* Subject under guardianship or trusteeship.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Change in optic nerve sheath diameter (ONSD) considered as an indirect marker for intracranial pressure (ICP) estimation | Baseline and five days of dry-immersion
  The optic nerve sheath diameter (ONSD) variations will be measured by echography.

SECONDARY OUTCOMES:
Change in the optic nerve fibers thickness | Baseline and five days of dry-immersion
  Thickness of the optic nerve fibers will be measured by Optical Coherence Tomography (OCT)
Change in cerebral structures and in venous circulation of the brain by MRI | Baseline and five days of dry-immersion
  Visualization of cerebral structures and intracranial venous system will be performed by MRI coupled with injection of gadolinium
Change in cerebral perfusion | Baseline and five days of dry-immersion
  Cerebral perfusion will be assessed by HMPAO scintigraphy
Change in intraocular pressure. | Baseline and five days of dry-immersion
  Intra ocular pressure (IOP) will be measured by applanation tonometry
Change in orthostatic tolerance | Baseline and five days of dry-immersion
  Orthostatic tolerance will be assessed during a Lower Body Negative Pressure test (LBNP test)
Change in body fluid compartments by bioelectrical impedance analysis | Baseline and during five days of dry-immersion
  Extracellular, intracellular and total body water will be estimated by bioimpedance
Change in circadian rhythms of blood pressure | Baseline and during the five days of the dry-immersion period
  Continuous 24-h recording of blood pressure will be performed by SOMNOtouch™ NIBP system designed for ambulatory continuous measurements
Measurement of the fluid shift towards the cephalic region by ultrasound | The first day to quantify the short term effect and the fourth day of dry-immersion to quantify the long term effect of fluid shift
  The hemodynamic and morphologic consequences of the fluid shift on the cephalic organs (thyroid, eyes), cephalic blood vessels (jugular vein, carotid, femoral, middle cerebral vein) will be investigated by ultrasound
Change of whole-body and skeletal muscle metabolic flexibility (i.e. capacity to adapt fuel oxidation to fuel availability) | Baseline and 4 days of dry-immersion
  Whole-body metabolic flexibility will be measured through the changes in respiratory quotient (RQ) from fasting state to postprandial state induced by high-carbohydrate standard meal, Skeletal muscle metabolic flexibility will be assessed in primary cell culture (cell isolation from biopsies of the vastus lateralis muscle).
Change in expression pattern of atrophic and phenotypic modifiers in skeletal muscle | Baseline and 5 days of dry-immersion
  Vastus Lateralis needle biopsies will be performed before and at the end of the 5 days of dry-immersion. The expression pattern of many proteins implied in the regulation of skeletal muscle homeostasis will be studied using biochemical technics.The contractile proteome will be investigated by analyzing the phenotype expression of myosin isoforms (heavy-MHC and light-MLC chains), regulatory proteins, i.e. troponin (TnI,TnC and TnT) and tropomyosin isoforms, main proteins implied in the sarcoplasmic reticulum function i.e. Ca-ATPase SERCA and Ca leakage channel RyR (primary antibodies from Sigma, Cell Signalling, Millipore).
Change in muscle transcriptome profile | Baseline and 5 days of dry-immersion
  Vastus Lateralis needle biopsies will be performed before and at the end of the 5 days of dry-immersion. The muscle gene expression will be analyzed by microarray technology
Measurement of muscle contractile properties using skinned fibers | Baseline and 5 days of dry-immersion
  Vastus Lateralis needle biopsies will be performed before and at the end of the 5 days of dry-immersion. Skinned fibers will be prepared by processing in skinning solution. Maximal tension and calcium affinity of single skinned fibers will be assessed using tensiometry.
Measurement of fat cell invasion into skeletal muscle | Baseline and 5 days of dry-immersion
  Vastus Lateralis needle biopsies will be performed before and at the end of the 5 days of dry-immersion. The expression of markers related to adipocytes structure and function (PPAR-γ, CEBP-α,CEBP-δ, lipoprotein lipase, ACLP, adipsin, leptin, adiponectin, FABP4, UCP1, IL6, IL15, CD36, GLUT4)will be quantified by RT-qPCR and western blotting. Additionally, the CD34+CD15+CD56- specific adipogenic progenitors of skeletal muscle will be quantified by RT-qPCR and western blotting.
Change in the balance of bone remodeling markers | Baseline, during and after 5 days of dry-immersion
  Concentration of bone formation markers [bone-specific Alkaline Phosphatase (bAP), procollagen type I N-terminal propeptide (P1NP), total osteocalcin, uncarboxylated and carboxylated osteocalcin] and of bone resorption markers [C-terminal cross-linked telopeptide of type I collagen (CTx)] will be analyzed by automated chemiluminescence immunoassay or by enzyme-immunoassay kits.
Change in the composition of the intervertebral disc (IVD). | Baseline and 5 days of dry-immersion
  The concentration of glycosaminoglycan (GAG) and water in the IVD will be measured by MRI with spectroscopy (MRS)

OTHER OUTCOMES:
Change in gut microbiota | Baseline, during and after 5 days of dry-immersion
  Shannon diversity and Simpson's indexes will be used as markers of microbial evenness and richness, respectively. Fresh fecal samples will be collected and frozen at -80°C. Bacterial DNA will be extracted, and then amplified by real-time PCR. 16S rRNA gene amplicons and Illumina HiSeq sequencing will be used to determine the diversity and structure comparisons of bacterial species. PCR amplifications will be sequenced and amplified using bioinformatics and biostatistics methods to obtain variations for different phylas and bacterial subfamily in each sample. Each individual will be compared to himself, and individual kinetics of gut microbiota changes will be performed.
Change in iron metabolism | Baseline, during and after 5 days of dry-immersion
  Transferrin saturation will be used as the best indicator of iron bioavailability. Circulating hepcidin level contributing to decrease transferrin saturation will also be measured.
Change in the contribution of visual and vestibular information used while performing mental transformations during a perspective-taking task. | Baseline, during and after 5 days of dry-immersion
  A perspective-taking task using virtual reality will be performed with concurrent recordings of eye-movements and cerebral metabolism. The drag-and-dropping the object will be recorded and concurrently physiological parameters (cerebral activity and gaze direction and duration).
Change in own-body representation. | Baseline, during and after 5 days of dry-immersion
  The following body parts will be measured on the real body of each participant (Total height, Head to left and right shoulder, Head to navel, Shoulder width, Upper and Lower arm length, Total arm length, Torso length, Navel to hip, Hip width, Upper and Lower leg length, Total leg length; limb and torso measures are performed left and right). We will also compute three ratios, torso length/hip width, arm length/shoulder width and leg length/hip width. All measures sill be entered into a program that draws the body shape.The computer program will then produce 13 body shapes that differ from 40% to 160% of the width of the original one, in 10% steps. A selection of 9 shapes out of the 13 is presented to the participant, ranked from the thinnest to the widest. All these measures and ratio will be compared to the corresponding real life measure (according to the scaling factor).

CONTACTS AND LOCATIONS:
Locations (1):
- Medes-Imps, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbeille P, Herault S, Fomina G, Roumy J, Alferova I, Gharib C. Influences of thigh cuffs on the cardiovascular system during 7-day head-down bed rest. J Appl Physiol (1985). 1999 Dec;87(6):2168-76. doi: 10.1152/jappl.1999.87.6.2168. PMID 10601164
- [Background] Balasubramanian S, Tepelus T, Stenger MB, Lee SMC, Laurie SS, Liu JHK, Feiveson AH, Sadda SR, Huang AS, Macias BR. Thigh Cuffs as a Countermeasure for Ocular Changes in Simulated Weightlessness. Ophthalmology. 2018 Mar;125(3):459-460. doi: 10.1016/j.ophtha.2017.10.023. Epub 2017 Nov 16. No abstract available. PMID 29153458
- [Background] De Abreu S, Amirova L, Murphy R, Wallace R, Twomey L, Gauquelin-Koch G, Raverot V, Larcher F, Custaud MA, Navasiolava N. Multi-System Deconditioning in 3-Day Dry Immersion without Daily Raise. Front Physiol. 2017 Oct 13;8:799. doi: 10.3389/fphys.2017.00799. eCollection 2017. PMID 29081752
- [Background] Kermorgant M, Leca F, Nasr N, Custaud MA, Geeraerts T, Czosnyka M, Arvanitis DN, Senard JM, Pavy-Le Traon A. Impacts of Simulated Weightlessness by Dry Immersion on Optic Nerve Sheath Diameter and Cerebral Autoregulation. Front Physiol. 2017 Oct 12;8:780. doi: 10.3389/fphys.2017.00780. eCollection 2017. PMID 29075198
- [Background] Navasiolava NM, Custaud MA, Tomilovskaya ES, Larina IM, Mano T, Gauquelin-Koch G, Gharib C, Kozlovskaya IB. Long-term dry immersion: review and prospects. Eur J Appl Physiol. 2011 Jul;111(7):1235-60. doi: 10.1007/s00421-010-1750-x. Epub 2010 Dec 14. PMID 21161267